CLINICAL TRIAL: NCT04064801
Title: Red Cell Distribution Width as a Predictor of Mortality in Acute Methanol Poisoning
Status: Completed | Type: Observational
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Barış Arslan, Adana City Training and Research Hospital, Adana Numune Training and Research Hospital
Other Study IDs: AdanaCTYHOSP
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Methanol Poisoning
Keywords: Alcohol, red blood cell distribution width, methanol poisoning, prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aimed to investigate the association between RDW and in-hospital mortality in methanol poisoning.

DETAILED DESCRIPTION:
RDW values have been found to be an independent predictor of the prognosis among patients with heart diseases, stroke,community-acquired pneumonia (CAP), pulmonary embolism, chronic obstructive pulmonary disease (COPD), septic shock, and acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

All patients aged ≥18 years who were admitted to emergency departments from January 2019 to January 2020 on account of acute methanol intoxication.

Exclusion Criteria:

Incomplete data, Malignancy, Severe anaemia, History of erythrocyte transfusion last 6 weeks

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute methanol toxicity who were diagnosed and treated at the Adana City Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | 7 day
Need for mechanical ventilation | 7 day

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No